CLINICAL TRIAL: NCT00003955
Title: A Phase II "Up-Front Window Study" of Irinotecan (CPT-11) Followed by Multimodal, Multiagent, Therapy for Selected Children and Adolescents With Newly Diagnosed Stage 4/Clinical Group IV Rhabdomyosarcoma: An IRS-V Study
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Metastatic Rhabdomyosarcoma or Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: D9802; COG-D9802 (Other: Children's Oncology Group); IRS-D9802 (Other: Intergroup Rhabdosarcoma Group); CCG-D9802 (Other: Children's Cancer Group); POG-D9802 (Other: Pediatric Oncology Group); CDR0000067154 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Sarcoma
Keywords: embryonal childhood rhabdomyosarcoma; alveolar childhood rhabdomyosarcoma; metastatic childhood soft tissue sarcoma; childhood malignant mesenchymoma; previously untreated childhood rhabdomyosarcoma; adult rhabdomyosarcoma; adult malignant mesenchymoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Malignant mesenchymal tumor; Rhabdomyosarcoma | interventions — Dactinomycin; Filgrastim; pegfilgrastim; sargramostim; Cyclophosphamide; Irinotecan; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: dactinomycin
Biological: filgrastim
Biological: pegfilgrastim
Biological: sargramostim
Drug: cyclophosphamide
Drug: irinotecan hydrochloride
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy combined with radiation therapy in treating patients who have metastatic rhabdomyosarcoma or sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with newly diagnosed high-risk metastatic stage IV/clinical group IV rhabdomyosarcoma treated with upfront window therapy comprising irinotecan and vincristine.
* Determine the toxic effects of this regimen in these patients.
* Determine the toxic effects of this regimen when given in alternating courses with vincristine, dactinomycin, and cyclophosphamide (VAC) as continuation therapy in patients with partial or complete response.
* Determine the overall and failure-free survival of patients treated with irinotecan and vincristine followed by VAC alone or VAC alternating with vincristine and irinotecan plus radiotherapy.
* Determine the pharmacokinetics of irinotecan and vincristine in these patients.

OUTLINE:

* Upfront window therapy: Patients receive vincristine IV on days 1 and 8 and irinotecan IV over 60 minutes on days 1-5 and 8-12. Treatment repeats every 21 days for a total of 2 courses. Patients experiencing partial or complete response proceed to regimen A. Patients experiencing stable or progressive disease proceed to regimen B.

  * Regimen A: Patients receive vincristine IV over 1 minute weekly on weeks 6-13, 15-19, 23-27, 29, 32-35, 38-39, and 41; dactinomycin IV over 1 minute weekly on weeks 6, 12, 23, 29, 35, and 41; and cyclophosphamide IV over 30-60 minutes weekly on weeks 6, 12, 16, 19, 23, 29, 35, and 41. Patients also receive irinotecan IV over 1 hour daily, 5 days a week, on weeks 9, 10, 26, 27, 32, 33, 38, and 39 and undergo radiotherapy daily, 5 days a week, on weeks 15-22.
  * Regimen B: Patients receive vincristine as in regimen A; dactinomycin IV over 1 minute weekly on weeks 6, 9, 12, 23, 26, 29, 32, 35, 38, and 41 and cyclophosphamide IV over 30-60 minutes weekly on weeks 6, 9, 12, 16, 19, 23, 26, 29, 32, 35, 38, and 41. Patients receive radiotherapy as in regimen A.

Patients who do not receive upfront window irinotecan/vincristine therapy are treated with standard therapy.

* Standard therapy: Patients receive vincristine IV over 1 minute weekly on weeks 0-13, 15-19, 23-27, 29, 32-35, 38, and 41; dactinomycin IV over 1 minute weekly on weeks 0, 6, 9, 12, 23, 26, 29, 32, 35, 38, and 41; and cyclophosphamide IV over 30-60 minutes weekly on weeks 0, 3, 6, 9, 12, 16, 19, 23, 26, 29, 32, 35, 38, and 41. Patients without evidence of intracranial extension receive radiotherapy once daily, 5 days a week, during weeks 15-22. Patients with evidence of intracranial extension, or who require emergency radiotherapy, receive radiotherapy during weeks 0-6. Dactinomycin is withheld during radiotherapy.

All patients receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously (SC) beginning 24 hours after completion of each course of chemotherapy and continuing until blood counts recover. Alternatively, patients may receive pegfilgrastim SC beginning 24-36 hours after completion of each course of chemotherapy and continuing until blood counts recover.

Patients are followed every 2 months for 1 year, every 4 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 18-46 patients will be accrued for this study within 9-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic stage IV/clinical group IV rhabdomyosarcoma, undifferentiated sarcoma, or ectomesenchymoma

  * No metastatic embryonal tumors in patients under 10 years of age, regardless of primary site
  * Metastatic tumors of parameningeal sites eligible
* Bidimensionally measurable disease
* No positive cerebrospinal fluid cytology or multiple intracranial metastases
* Patients presenting with the following are only eligible for continuation therapy and may not receive irinotecan/vincristine upfront window therapy:

  * Evidence of base of skull erosion or skull metastatic disease that displaces or indents the dura, compresses the brain parenchyma, or causes evidence of cranial nerve palsy
  * Tumor that touches or displaces the spinal cord
  * Evidence of intracranial primary tumor extension
  * Tumors that could cause potentially life-threatening complications (e.g., renal, airway) with progression due to location and/or growth rate
  * Requires emergency radiotherapy
  * Lab values are consistent with disseminated intravascular coagulation

PATIENT CHARACTERISTICS:

Age:

* Under 50 (alveolar rhabdomyosarcoma, undifferentiated sarcoma, and ectomesenchymoma patients)
* 10 to 49 (embryonal histology patients)

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count greater than 1,000/mm^3*
* Platelet count greater than 150,000/mm^3* NOTE: *Unless there is tumor involvement of bone marrow

Hepatic:

* Bilirubin less than 1.5 mg/dL
* PT, PTT, and fibrinogen less than 1.5 times upper limit of normal

Renal:

* Creatinine less than 1.2 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior steroids allowed

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy

Surgery:

* No more than 42 days since prior initial surgical procedure, including biopsy for diagnosis

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 1999-09; Primary Completion 2005-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Alberto S. Pappo, MD, Study Chair — Texas Children's Cancer Center
Locations (237):
- United States (209):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center, San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - University of Connecticut Comprehensive Cancer Center at University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics - Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Comprehensive Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital at University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Puerto Rico (2):
  - Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Soft Tissue Sarcoma Committee of the Children's Oncology Group; Lager JJ, Lyden ER, Anderson JR, Pappo AS, Meyer WH, Breitfeld PP. Pooled analysis of phase II window studies in children with contemporary high-risk metastatic rhabdomyosarcoma: a report from the Soft Tissue Sarcoma Committee of the Children's Oncology Group. J Clin Oncol. 2006 Jul 20;24(21):3415-22. doi: 10.1200/JCO.2005.01.9497. PMID 16849756
- [Result] Pappo AS, Lyden E, Breitfeld P, Donaldson SS, Wiener E, Parham D, Crews KR, Houghton P, Meyer WH; Children's Oncology Group. Two consecutive phase II window trials of irinotecan alone or in combination with vincristine for the treatment of metastatic rhabdomyosarcoma: the Children's Oncology Group. J Clin Oncol. 2007 Feb 1;25(4):362-9. doi: 10.1200/JCO.2006.07.1720. PMID 17264331